CLINICAL TRIAL: NCT00186316
Title: A Phase I/II Study of Vaccine Therapy for Multiple Myeloma Utilizing Idiotype-Pulsed Allogeneic Dendritic Cells
Brief Title: Vaccine Therapy for Multiple Myeloma Utilizing Idiotype-Pulsed Allogeneic Dendritic Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald Levy, Principal Investigator, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT155; 79000; BMT155; NCT00186316
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Biological: Idiotype-pulsed allogeneic dendritic cells

SUMMARY:
Patients with Multiple myeloma who have undergone non-myeloablative allogeneic stem cell transplant will receive 6 vaccinations of donor derived dendritic cells combined with specific protein produced by multiple myeloma.

DETAILED DESCRIPTION:
To evaluate feasibility and safety of vaccination with allogeneic idiotype-pulsed dendritic cells following mixed chimeric allogeneic transplantation for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:1. For specimen collection and idiotype protein development:

* Must be secretory myeloma with at least .5g/dl serum IgG protein
* Clinically stage 2 or 3 multiple myeloma
* Karnofsky performance status of 70 or greater

  2. For Vaccination:
* Eligible patients must have completed tandem autologous and nonmyeloablative allogeneic transplant for multiple myeloma at Stanford University Medical Center with stable disease or complete response to prevaccine therapy
* Karnofsky performance status of 70 or greater.
* ALT and AST must be <2X upper limit of normal. Total bilirubin < 1.5X upper limit of normal.
* Serum creatinine <1.5X upper limit of normal.
* Hemoglobin >9g/dl
* Patients must be HIV negative.
* Patients must provide signed, informed consent

Donor Inclusion Criteria (allo donor is the same donor used for non-myeloablative transplant)

* Age >17 years
* HIV negative
* Must provide signed, informed consent Exclusion Criteria:1. For specimen collection and idiotype protein development:
* Patients with non-secretory myeloma
* Severe psychological or medical illness
* Pregnant or lactating women
* Subjects with > Grade I toxicity by NCI-CTC v 3.0
* Subjects with prognosis < 6 months

  2. For Vaccination:
* < 75 mg of idiotype protein purified from the patients serum
* < 25 million allogeneic idiotype-pulsed dendritic cells produced for vaccination
* Evidence of grade II-IV acute GVHD (defined in section 5E)
* Patients with evidence of myeloma disease progression as (defined below)
* Severe psychological or medical illness or concomitant medications which may interfere with the study as determined by the clinical investigator
* Patients on any other investigational agents
* Pregnant or lactating women
* Patients on any therapy for multiple myeloma or any chemotherapy drug, or immunomodulatory agent for treatment of multiple myeloma (e.g. thalidomide)
* Any patient on more than two of the following immunosuppressive agents or at a dose greater than that indicated for a single immunosuppressive agent:

  1. Mycophenolate Mofetil (MMF)- no greater than 1000mg twice a day
  2. Prednisone- no greater than .5mg/kg/day
  3. Cyclosporine- no greater than 300mg/day
  4. Tacrolimus (FK506)- no greater than 4mg/day

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Patient will complete 4 vaccinations of monthly interval

SECONDARY OUTCOMES:
Evaluation of immune response. Immune response analysis will be done on all patients who are enrolled in the study. Patients who completed a minimum of 4 vaccinations will be included in immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States